CLINICAL TRIAL: NCT04893278
Title: Use of Virtual Reality as An Adjunct for Anesthesia During Procedures in the Electrophysiology Laboratory: A Pilot and Feasibility Study
Brief Title: Virtual Reality in Electrophysiology Laboratory (EP)
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Klaus D. Torp, Principal Investigator, Mayo Clinic
Other Study IDs: 21-002644
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: PVC - Premature Ventricular Complex; Ablation
Keywords: virtual reality
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Virtual reality
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — Use of Virtual reality goggles during procedure

SUMMARY:
The purpose of this study is to evaluate the use of virtual reality (VR) technology as adjunct to routine anesthesia care for patients undergoing electrophysiology (EP) procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients scheduled for electrophysiology procedure with MAC.
* Subject willing to participate and able to provide informed consent.

Exclusion Criteria:

* Age < 18 years old.
* History of motion sickness or blindness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from patients undergoing procedures under monitored anesthesia care.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Virtual reality as distractor | Up to 2hours
  Evaluate patients' experience and satisfaction with using virutal reality during electrophysiology procedures

SECONDARY OUTCOMES:
Impact of virtual reality use on pharmacological therapy | Up to 2 hours
  Evalute the amount of medications use during the procedure
Impact of virtual reality on electrophysilogy procedure | Up to 2 hours
  Evaluate success rate of completing ablation while patient is utilizing virtual reality

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Torp, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials